CLINICAL TRIAL: NCT00770978
Title: Open-Label, Parallel Group, Multiple-dose Study of Ceftobiprole to Evaluate the Plasma Pharmacokinetics in Adults in Intensive Care Units
Brief Title: Open Label Study of Ceftobiprole to Evaluate Pharmacokinetics in Adults Hospitalized in the ICU
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Basilea Pharmaceutica (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR014911; NOS-1001 (Other: Basilea Internal Reference)
Record Dates: First submitted 2008-10-09; First posted 2008-10-10 (Estimated); Last update posted 2012-07-30 (Estimated); Status verified 2012-07

CONDITIONS: ICU
Keywords: ICU

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ceftobiprole q12h (Experimental): Ceftobiprole, 1G q12h as 4 hour infusions, on Day 1 and Ceftobiprole, 1G as single 4 hour infusion on Day 2
  Interventions: Drug: ceftobiprole q12h
- Ceftobiprole q8h (Experimental): Ceftobiprole, 1G q8h as 4 hour infusions, on Day 1 and Ceftobiprole, 1G as single 4 hour infusion on Day 2
  Interventions: Drug: ceftobiprole q8h

INTERVENTIONS:
Drug: ceftobiprole q12h — Ceftobiprole, 1G q12h as 4 hour infusions, on Day 1 and Ceftobiprole, 1G as single 4 hour infusion on Day 2
  Arms: Ceftobiprole q12h
Drug: ceftobiprole q8h — Ceftobiprole, 1G q8h as 4 hour infusions, on Day 1 and Ceftobiprole, 1G as single 4 hour infusion on Day 2
  Arms: Ceftobiprole q8h

SUMMARY:
The purpose of this research study is to measure the levels of ceftobiprole in the blood and urine during and after administration of four doses of ceftobiprole. Safety of the drug will also be evaluated.

DETAILED DESCRIPTION:
Patients will receive an intravenous dose of ceftobiprole infused over 4 hours. Multiple blood samples will be obtained to determine the concentration of ceftobiprole in the plasma. Pharmacokinetic parameters such as clearance and volume of distribution will be calculated. 1000mg every 8hours or every 12 hours

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent
* Between 18 and 75 years of age inclusive
* BMI 18 - 35 inclusive
* Albumin < 3.3 g/dL or clinical evidence of edema
* Negative Pregnancy test
* Expected survival of at least 7 days

Exclusion Criteria:

* Known drug allergy (including penicillin, cephalosporin, carbapenems, or other beta-lactams)
* Renal impairment (CrCl < 50 mL/min) or dialysis
* History of seizures
* ALT or AST > 5 times upper normal limit
* Sustained shock, unresponsive to sympathomimetics
* Conditions that may have jeopardized adherence to the protocol (NYHA Class 4 cardiac disease, >15% total body burn or significant third degree burn)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2008-11; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (to measure the levels of ceftobiprole in the blood and urine) during dosing and 24 hours after last dose | 3 days

SECONDARY OUTCOMES:
Safety will be evaluated throughout the study. | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (13):
- United States (4):
  - Birmingham, Alabama
  - Chicago, Illinois
  - Beech Grove, Indiana
  - Omaha, Nebraska
- Belgium (2):
  - Aalst
  - Edegem
- Greenfield Park, Quebec, Canada
- Jerusalem, Israel
- South Korea (3):
  - Gwangju
  - Incheon
  - Seoul
- Spain (2):
  - Barcelona
  - Madrid